CLINICAL TRIAL: NCT02501408
Title: Comparaison du Pied Bionique Proprio-Foot® Versus le Pied Habituel Chez Les amputés Tibiaux
Brief Title: Comparing New Prothesis PROPRIO-FOOT® Versus Usual Prothesis Tasks Tibial Amputees
Acronym: PROPRIO-FOOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00374-43
Record Dates: First submitted 2015-07-16; First posted 2015-07-17 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2016-12

CONDITIONS: Lower Limb Amputation at Ankle (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propriofoot prosthesis (Experimental): New propriofoot prosthesis is worn instead of usual prosthesis foer 1 month
  Interventions: Device: propriofoot prosthesis
- Control (No Intervention): Usual prosthesis is worn for 1 month

INTERVENTIONS:
Device: propriofoot prosthesis — Adaptation of the device and evaluation after 1 month at home using the studied device
  Arms: Propriofoot prosthesis

SUMMARY:
Evaluate a new porosthetic device in lower limb amputees.

DETAILED DESCRIPTION:
Randomisation between usual and new prosthesis Cross over study of walking performance and VO2 on treadmill with the two devices after 1 month adaptation to each system.

ELIGIBILITY:
Inclusion Criteria:

* Tibial amputation
* Ability top walk on treadmill
* Stable prosthesis for at least 3 months

Exclusion Criteria:

* Bilateral amputation
* Cancer
* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
oxygen consumption | 1 mois after adpatation of the selected device
  Measurement on treadmill

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Abraham, Principal Investigator — University Hospital, Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France